CLINICAL TRIAL: NCT06193850
Title: Observational Study on the Quality of Life of Patients Attending General Urology, Sexual Medicine, Reproductive Medicine, Uro-oncology, Neuro-urology, Functional Urology Clinics
Brief Title: Protocol N. 2014 - Observational Study on the Quality of Life of Outpatients
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: 2014 Ambulatoriali
Record Dates: First submitted 2023-11-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Urologic Diseases; Male Infertility; Sexual Medicine
Keywords: Male Infertility; urology; rare male cancer
MeSH Terms: conditions — Urologic Diseases; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uro-andrologic patients: Subjects belonging to general urology, sexual medicine, reproductive medicine, functional urology, neuro-urology and uro-oncology clinics.
  Interventions: Other: Observation during time

INTERVENTIONS:
Other: Observation during time — Evaluation through clinical investigation and questionnaires useful for evaluating the patient's psycho-physical conditions

SUMMARY:
Prospective observational study on the quality of life of patients attending general urology, sexual medicine, reproductive medicine, functional urology, neuro-urology and uro-oncology clinics.The data relating to the clinical conditions (disease state, psychological and related to quality of life) of the patients belonging to the above-mentioned clinics will be collected in a specially designed database which will allow us to extract the data in a simple and safe way used for statistical analyses. in clinical research.

DETAILED DESCRIPTION:
The Department of Urology has been engaged for years in the field of medical and surgical research relating to benign and oncological pathologies of the prostate, kidney, excretory tract, testicle, as well as urinary continence and dysfunctions of the sexual and reproductive sphere. The accurate acquisition of clinical and psychometric data before and after any treatment, the follow-up analysis, the attention to the patient's global quality of life (QoL) in relation to the particular organic functions affected by the disease, are at the basis of all the medical advances that can be achieved to guarantee ever better care of the individual's health. In the context of urological clinical practice, outpatient activity plays a fundamental role. This activity, which ranges from general urology to sexual medicine, reproductive medicine, functional urology, neuro-urology and uro-oncology, allows us to come into contact with a large number of patients suffering from the most common uropathologies -andrological .

Numerous studies have demonstrated how the treatment and outpatient management of such patients significantly impacts not only the underlying pathology but also their quality of life.

The outpatient management of the urological patient ranges from the recognition of the basic pathology to the diagnosis through the request for clinical-laboratory-instrumental investigations, to the possible indication for a medical or surgical treatment and to the follow-up of the patient.

The main objectives of this data archive are:

1. Collect clinical, instrumental, laboratory, psychometric and sociodemographic data in patients suffering from a uro-andrological pathology who require a consultation in one of the clinics mentioned above.
2. Collect data on the natural history of the pathologies in question and on the patients' quality of life in order to analyze the predictive factors of persistence and recurrence of symptoms, improvement or worsening of the clinical picture, and possible progression of the disease (both in benign and malignant form) and improve the care and treatment of the patients under examination.
3. Having a follow-up and related studies with a number and above all an extension over time that, to date, is not present in the literature or in any scientific production.

ELIGIBILITY:
Inclusion Criteria:

* subjects belonging to general urology, sexual medicine, reproductive medicine, functional urology, neuro-urology and uro-oncology clinics.
* subjects >= 18 years old
* signature of informed consent

Exclusion Criteria:

* - subjects < 18 years
* presence of mental or physical disability that may prevent the patient from answering the questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population of interest is characterised by: patients who came for outpatient visits to the general urology, sexual medicine, reproductive medicine, functional urology, neuro-urology and uro-oncology clinics.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-02-24 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2045-01-31 (Estimated)

PRIMARY OUTCOMES:
Sexual function - Erectile Function | Baseline and up to 6 months
  Sexual function investigated through: "International Index of Erectile Function" questionnaire IIEF (scoring: 1 - 30 - 6-10: severe; 11-16: Moderate; 17-25: mild; 26-30: absence);
Sexual function - premature ejaculation | Baseline and up to 6 months
  Premature ejaculation investigated through PEDT questionnaire (; Scoring: 0 - 20. <=8 absence; 9-10 probable; >=11 premature ejaculation);
Sexual function - male sexual health | Baseline and up to 6 months
  Male sexual health investigated through MSHQ questionnaire (25-item, range: 7 - 80, greater score indicating better function and through Androtest (1 - 32; > 8 = out of the norm);
Sexual function - androgen deficiency | Baseline and up to 6 months
  Androgen deficiency in elderly males investigated through ADAM questionnaire (range 10 - 50, 10 = absence and 50 = maximal,
Sexual function - satisfaction with treatment of erection problems | Baseline and up to 6 months
  satisfaction with treatment of erection problems investigated through EDITS questionnaire (range = 0-100; higher scores =more treatment satisfaction),
Female sexual function | Baseline and up to 6 months
  Female sexual function investigated through "Female Sexual Function Index" questionnaire - FSFI (range 2 - 36, lower scores = worse sexual functioning),;
Sexual function - sexual distress | Baseline and up to 6 months
  Sexual distress investigated through "Sexual Distress Scale" questionnaire - SDS (range 12- 48, sexual distress = > 15).

SECONDARY OUTCOMES:
Prostate function - Prostatic Symptoms | Baseline and up to 6 months
  Prostatic Symptoms investigated through IPSS questionnaire "International Prostatic Symptoms Score": , Scoring 0 -7, 0-7 mild symptoms, 8-19 moderate symptoms, 20-35 severe symptoms
Psychological state | Baseline and up to 6 months
  Psychological state investigated through Beck Beck Depression Inventory: Range score 1 - 63; 1-10: normal; 11-16: Mild mood disturbance; 17-20: Borderline clinical depression; 21-30: Moderate depression; 31-40: Severe depression; over 40: Extreme depression.
Prostate function - Incontinence Questionnaire | Baseline and up to 6 months
  Incontinence Questionnaire investigated through ICIQ-SF questionnaire (maximum score of 21; the higher the score, the more severe is the UI, but there is no normal score)
Overactive Bladder | Baseline and up to 6 months
  Overactive Bladder investigated through OAB-q - Overactive Bladder Questionnaire: the score for each of OAB-q domain are summed and transformed to a score ranging from zero to 100. Higher scores indicate more severe symptoms or better quality of life.
Prostate function | Baseline and up to 6 months
  Prostate function investigated through National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) questionnaire: total score range from 0 to 43, three subscales addressing pain (score range 0-21), urinary symptoms (score range 0-10), and quality of life (QOL) (score range 0-12)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy